CLINICAL TRIAL: NCT03413839
Title: Physiotherapeutic Scoliosis Specific Exercises As Treatment for Adult Degenerative Scoliosis vs Conventional Physical Therapy Exercises
Brief Title: Physiotherapeutic Scoliosis Specific Exercises As Treatment for Adult Degenerative Scoliosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No research resources to complete study
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAQ9761
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Degenerative Scoliosis
Keywords: Scoliosis; PSSE
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSSE Group (Experimental): Individuals will receive at least 6 sessions of physiotherapeutic scoliosis specific exercises (PSSE) (Schroth) physical therapy. Patients will also be required to perform exercises 5x/wk for 15 minutes at home. Compliance will be monitored by written log and weekly phone check-in after 8 weeks.
  Interventions: Behavioral: Physiotherapeutic Scoliosis Specific Exercises (PSSE)
- Conventional PT Group (Other): Individuals will receive at least 6 sessions of conventional physical therapy (PT). Patients will also be required to perform exercises 5x/wk for 15 minutes at home. Compliance will be monitored by written log and weekly phone check-in after 8 weeks.
  Interventions: Behavioral: Conventional Physical Therapy (PT)

INTERVENTIONS:
Behavioral: Physiotherapeutic Scoliosis Specific Exercises (PSSE) — Exercises with emphasis on trunk extensor strengthening, and teaching patient better postural strategies in supine, sidelying, sitting, standing, and dynamic movements (walking, squatting), led by a PSSE-trained physical therapist.
  Other Names: PSSE
  Arms: PSSE Group
Behavioral: Conventional Physical Therapy (PT) — Conventional PT includes generalized pelvis, and trunk strengthening, lower extremity (LE) stretching, and use of modalities (ice and heat), iontophoresis and E-Stim.
  Arms: Conventional PT Group

SUMMARY:
This is a pilot study to lead to a larger prospective, randomized, controlled study of older adult (ages 50 and older) spinal patients with thoracolumbar/lumbar scoliosis evaluating improvement with physiotherapeutic scoliosis-specific exercise (PSSE) compared to traditional low back physical therapy (PT).

DETAILED DESCRIPTION:
Adult scoliosis with chronic back pain is a very complex condition. Chronic back pain remains one of our country's most costly conditions to manage and treat. Many of these patients have difficulty with activities of daily living (ADL), household and community ambulation, and maintaining their professional career. The intervention options for this population remain limited, with surgery being the only one that has shown improvements in health related quality of life and an overall decrease in the complaints of pain. However, the costs of surgery and additional complications are limitations to this treatment option.There has been increased attention and interest in the medical community looking at the effects of Physiotherapeutic Scoliosis Specific Exercises (PSSE) on curve progression, improvements in health related quality of life, and pain. The investigators hypothesize that PSSE can directly affect radiological parameters, such as the sagittal vertical axis (SVA), as well as showing improvements in health related quality of life using subjective patient specific outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years old
* Diagnosis of adolescent idiopathic scoliosis or adult idiopathic scoliosis; either with a Cobb angle ranging from 20-100 degrees
* Complaint of back pain that has lasted longer than 6 weeks

Exclusion Criteria:

* Any patient who has completed PSSE in the past
* Previous spinal surgery, trauma, or presence of neoplasms
* Diagnosis of congenital or neuromuscular scoliosis
* Subjects who are involved in concurrent interventions other than conventional physical therapy (PT)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Score for Back Pain | Up to 2 years
  The VAS is a psychometric response scale which measures subjective characteristics or attitudes that cannot be directly measured. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Score on Scoliosis Research Society 22-item (SRS-22r) | Up to 6 months
  Outcome measure designed by the Scoliosis Research Society that is specially designed for patients with scoliosis and evaluates their scores for self-image, pain, mental health, and function. It contained 22 items contributing to five main domains: Function (5 items), Pain (5 items), Self-image/appearance (5 items), Mental Health (5 items), Satisfaction with Treatment (Current/Previously performed-2 items). Scores range from 5 (best) to 1 (worst).
Score on Oswestry Disability Index (ODI) | Up to 6 months
  The ODI is a self-completed questionnaire containing 10 topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Chen, MD, MPH, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bess S, Schwab F, Lafage V, Shaffrey CI, Ames CP. Classifications for adult spinal deformity and use of the Scoliosis Research Society-Schwab Adult Spinal Deformity Classification. Neurosurg Clin N Am. 2013 Apr;24(2):185-93. doi: 10.1016/j.nec.2012.12.008. PMID 23561557
- [Background] Li G, Passias P, Kozanek M, Fu E, Wang S, Xia Q, Li G, Rand FE, Wood KB. Adult scoliosis in patients over sixty-five years of age: outcomes of operative versus nonoperative treatment at a minimum two-year follow-up. Spine (Phila Pa 1976). 2009 Sep 15;34(20):2165-70. doi: 10.1097/BRS.0b013e3181b3ff0c. PMID 19713875
- [Background] Monticone M, Ambrosini E, Cazzaniga D, Rocca B, Motta L, Cerri C, Brayda-Bruno M, Lovi A. Adults with idiopathic scoliosis improve disability after motor and cognitive rehabilitation: results of a randomised controlled trial. Eur Spine J. 2016 Oct;25(10):3120-3129. doi: 10.1007/s00586-016-4528-y. Epub 2016 Mar 25. PMID 27015689
- [Background] Bridwell KH, Glassman S, Horton W, Shaffrey C, Schwab F, Zebala LP, Lenke LG, Hilton JF, Shainline M, Baldus C, Wootten D. Does treatment (nonoperative and operative) improve the two-year quality of life in patients with adult symptomatic lumbar scoliosis: a prospective multicenter evidence-based medicine study. Spine (Phila Pa 1976). 2009 Sep 15;34(20):2171-8. doi: 10.1097/BRS.0b013e3181a8fdc8. PMID 19752703
- [Background] Weinstein JN, Lurie JD, Tosteson TD, Zhao W, Blood EA, Tosteson AN, Birkmeyer N, Herkowitz H, Longley M, Lenke L, Emery S, Hu SS. Surgical compared with nonoperative treatment for lumbar degenerative spondylolisthesis. four-year results in the Spine Patient Outcomes Research Trial (SPORT) randomized and observational cohorts. J Bone Joint Surg Am. 2009 Jun;91(6):1295-304. doi: 10.2106/JBJS.H.00913. PMID 19487505
- [Background] Weinstein JN, Lurie JD, Tosteson TD, Hanscom B, Tosteson AN, Blood EA, Birkmeyer NJ, Hilibrand AS, Herkowitz H, Cammisa FP, Albert TJ, Emery SE, Lenke LG, Abdu WA, Longley M, Errico TJ, Hu SS. Surgical versus nonsurgical treatment for lumbar degenerative spondylolisthesis. N Engl J Med. 2007 May 31;356(22):2257-70. doi: 10.1056/NEJMoa070302. PMID 17538085
- [Background] Schwab F, Dubey A, Gamez L, El Fegoun AB, Hwang K, Pagala M, Farcy JP. Adult scoliosis: prevalence, SF-36, and nutritional parameters in an elderly volunteer population. Spine (Phila Pa 1976). 2005 May 1;30(9):1082-5. doi: 10.1097/01.brs.0000160842.43482.cd. PMID 15864163
- [Background] Kuru T, Yeldan I, Dereli EE, Ozdincler AR, Dikici F, Colak I. The efficacy of three-dimensional Schroth exercises in adolescent idiopathic scoliosis: a randomised controlled clinical trial. Clin Rehabil. 2016 Feb;30(2):181-90. doi: 10.1177/0269215515575745. Epub 2015 Mar 16. PMID 25780260
- [Background] Negrini A, Negrini MG, Donzelli S, Romano M, Zaina F, Negrini S. Scoliosis-Specific exercises can reduce the progression of severe curves in adult idiopathic scoliosis: a long-term cohort study. Scoliosis. 2015 Jul 11;10:20. doi: 10.1186/s13013-015-0044-9. eCollection 2015. PMID 26279670
- [Background] Negrini S, Donzelli S, Lusini M, Minnella S, Zaina F. The effectiveness of combined bracing and exercise in adolescent idiopathic scoliosis based on SRS and SOSORT criteria: a prospective study. BMC Musculoskelet Disord. 2014 Aug 6;15:263. doi: 10.1186/1471-2474-15-263. PMID 25095800